CLINICAL TRIAL: NCT03355313
Title: Use of Low-level Laser Therapy on Children Aged One to Five Years With Energy-protein Malnutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, PROFESOR, University of Nove de Julho
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Malnutrition
Record Dates: First submitted 2017-11-07; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Malnutrition, Child
Keywords: saliva; Low-level light therapy; salivary glands
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Nutritional status of 50 children will be measured according the World Health Organization. The volume of saliva will be measured and, also, the salivary flow rate(mL/min) and buffering capacity will be determined. Concentrations of salivary IgA in all samples will be measured using a ELISA kit. Laser will be administered for 10 seconds on four intraoral points and four extraoral points in the region of the parotid glands bilaterally as well as one intraoral point and one extraoral point in the regions of the submandibular and sublingual glands. Three sessions of laser therapy will occur (after the collection of saliva, 7 and 14 days after the first session, respectively). The final saliva collection will be performed after the third laser session. The laser will be adjusted according to the following parameters: 808nm, 4 J, Continuous and contact mode,100mW, Irradiation at target (mW/cm2)=2500,Irradiated area (cm2)=0.40.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low level light therapy 1 (Experimental)
  Interventions: Radiation: Low level Light therapy
- Low level light therapy 2 (Experimental)
  Interventions: Radiation: Low level Light therapy
- Low level light therapy 3 (Experimental)
  Interventions: Radiation: Low level Light therapy

INTERVENTIONS:
Radiation: Low level Light therapy — Laser will be administered for 10 seconds on four intraoral points and four extraoral points in the region of the parotid glands bilaterally as well as one intraoral point and one extraoral point in the regions of the submandibular and sublingual glands.

SUMMARY:
Malnutrition is a clinical-social disease caused by multiple prenatal, intrauterine and postnatal factors as well as social, political and cultural determinants (distal causes). Despite the global and national reductions in the number of cases, malnutrition continues to be a public health problem, with greater prevalence in pockets of poverty found in the northern and northeastern regions of Brazil.

Episodes of malnutrition in early childhood, with consequent calcium, phosphate and vitamin A, C and D deficiencies, can increase one's susceptibility to dental caries through three probable mechanisms: defects in tooth formation (odontogenesis), delayed tooth eruption and alterations in the salivary glands.

It is likely that the significant increase in susceptibility to caries in malnourished individuals stems from alterations in the salivary secretion rate, since a reduction in salivary flow (salivary gland atrophy) increases the susceptibility to both dental caries and dental erosion. As saliva is the main defense factor of the oral cavity, a reduction/change in its physical properties (secretion rate and buffering capacity) can cause immunological disorders that affect an individual's defense capacity.

Studies have demonstrated that salivary immunoglobulin A (IgA) also plays an important role in the immunity of the oral mucosa. Indeed, patients with IgA deficiency can experience recurring upper airway (tonsillitis, ear infection and sinusitis), lower airway (pneumonia) and gastrointestinal (diarrhea and parasitosis) infections.

The investigation of mechanisms that can reduce the impact of malnutrition on the defenses of the organism is of the utmost important and interest to public health. Among such mechanisms, low-level laser therapy has demonstrated effectiveness in the treatment of diverse conditions and disease through the promotion of the biomodulation of the cell metabolism and due to its analgesic and anti-inflammatory properties with no mutagenic or photothermal effects.

DETAILED DESCRIPTION:
Laser stimulation of the major salivary glands to produce more saliva occurs through the increase in local circulation due to vasodilatation, the induction of the proliferation of glandular cells and cell respiration/ATP (adenosine triphosphate) synthesis as well as the release of growth factors and cytokines to stimulate protein exocytosis. With regard to an increase in salivary IgA, low-level laser intensifies the activation of B lymphocytes, which differentiate into plasma cells, thereby contributing to the increase in immunoglobulin levels.

The study of salivary aspects in malnourished children and possible treatments that can be used to improve salivary quality and quantity in these children has significant social relevance, as saliva is one of the main mechanisms against infection and participates in essential functions of life, such as swallowing and the maintenance of oral health.

An experimental cross-sectional study is proposed, which will be conducted at the Center for Educational and Nutrition Recovery in the city of Maceió, state of Alagoas, Brazil, and University Nove de Julho (UNINOVE) in the city of Sao Paulo, Brazil. This project has been approved by CESMAC ethics committee (CAAE 71961317.1.0000.0039).

ELIGIBILITY:
Inclusion Criteria:

* Children aged one to five years enrolled at the Center for Educational and Nutrition Recovery in the city of Maceió whose parent/guardians signed as statement of informed consent agreeing to the participation of the children.
* Children suffering of malnutrition.

Exclusion Criteria:

* Children aged one to five years not enrolled at the Center for Educational and Nutrition Recovery in the city of Maceió and children whose parents/guardians did not sign a statement of informed consent.
* Children not suffering of malnutrition.

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Low-level laser irradiation on the salivary glands | 3 weeks
  Laser will be administered for 10 seconds on four intraoral points and four extraoral points in the region of the parotid glands bilaterally as well as one intraoral point and one extraoral point in the regions of the submandibular and sublingual glands.
  The laser will be adjusted according to the following parameters:
  Central wavelength (nm)= 808, Spectral band width (FWHM) (nm)= 2, Operational mode= Continuous, Mean radiant power (mW)=100, Polarization= Randomized, Aperture diameter (cm) =0.2, Irradiation at aperture (mW/cm2)= 2500, Beam profile= Multimodal, Beam spot on target (cm2)= 0.04, Irradiation at target (mW/cm2)= 2500, Exposure time (s)= 40, Radiant exposure (J/cm2)=100.0, Radiant energy (J)= 4, Number of points irradiated=10, Irradiated area (cm2) =0.40, Application method= Contact, Number of treatment sessions= 3, Frequency of treatment sessions per week =1, Total radiant energy (J) =40.

SECONDARY OUTCOMES:
Length/Height | 1 week
  Length - A wooden measuring board (also called sliding board) will be used for measuring the length of children under two years old to the nearest millimetre.
  Height - This is measured with the child in a standing position.
Weight | 1 week
  A weighing sling (spring balance), also called the 'Salter Scale' will be used for measuring the weight of children under two years old, to the nearest 0.1 kg. Children over two years a beam balance will be used and the measurement is also to the nearest 0.1 kg.
Saliva flow rate measurement | 3 weeks
  Salivary flow rates can be reduced significantly in individuals who have suffered severe malnutrition in early childhood.
  Saliva parameters of children with malnutrition will be measured and compared to normal values.
  Total resting saliva will be collected between 9 and 11 am (to avoid the influence of circadian rhythm) using the drainage method.
  The child will be instructed to swallow prior to the collection and then instructed not to swallow, allowing the saliva to drain between the lips (which will be separated) into a test tube (aspirator) connected to a 15-mL Flacon tube positioned near the mouth.
  Collection time will be five minutes. The volume of saliva will be measured and the salivary flow rate will be determined (mL/min).
  Normal unstimulated salivary flux is above 0,2 ml/min. This measure was done in the samples of saliva before and after the lasertherapy for all patients.
Buffering Capacity of saliva | 3 weeks
  One aliquot (1 ml) of saliva will be transferred immediately to a small tube (capacity: 5 ml) for titration with hydrochloric acid 0.005 Ne. The tube will be shaken for 15 seconds and buffering capacity will be measured using a glass electrode (Orion) coupled to a pH meter.
  The reading of this test is performed based on the following parameters: pH 3.0 to 4.0 = very low to low buffering capacity; pH 4.5 to 5.0 = intermediate buffering capacity; and pH ≥ 5.5 = normal/good buffering capacity.
  This measure was done in the samples of saliva before and after the lasertherapy for all patients.
Analysis of salivary IgA | 3 weeks
  Concentrations of salivary IgA in all samples will be measured using a commercial enzyme-linked immunosorbent assay (ELISA) kit.
  Salivary IgA (µg/ml) in each sample will be calculated using a standard curve obtained from the calibrators in the kit.
  Normal saliva in children from 12 to 23 months = 2.3 ± 1.5 (mg/dl) Normal saliva in children from 24 to 71 months = 4.1 ± 2.4 (mg/dl) This measure was done in the samples of saliva before and after the lasertherapy for all patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Centro de Educação e Recuperação Nutricional, Maceió, Alagoas
  - University of Nove de Julho, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] Johansson I, Saellstrom AK, Rajan BP, Parameswaran A. Salivary flow and dental caries in Indian children suffering from chronic malnutrition. Caries Res. 1992;26(1):38-43. doi: 10.1159/000261425. PMID 1568235
- [Background] Vidovic Juras D, Lukac J, Cekic-Arambasin A, Vidovic A, Canjuga I, Sikora M, Carek A, Ledinsky M. Effects of low-level laser treatment on mouth dryness. Coll Antropol. 2010 Sep;34(3):1039-43. PMID 20977100
- [Background] Loncar B, Stipetic MM, Baricevic M, Risovic D. The effect of low-level laser therapy on salivary glands in patients with xerostomia. Photomed Laser Surg. 2011 Mar;29(3):171-5. doi: 10.1089/pho.2010.2792. Epub 2010 Nov 6. PMID 21054200
- [Background] Michalke B, Rossbach B, Goen T, Schaferhenrich A, Scherer G. Saliva as a matrix for human biomonitoring in occupational and environmental medicine. Int Arch Occup Environ Health. 2015 Jan;88(1):1-44. doi: 10.1007/s00420-014-0938-5. Epub 2014 Mar 12. PMID 24619390
- [Background] Navazesh M, Christensen CM. A comparison of whole mouth resting and stimulated salivary measurement procedures. J Dent Res. 1982 Oct;61(10):1158-62. doi: 10.1177/00220345820610100901. No abstract available. PMID 6956596
- [Background] Psoter WJ, Spielman AL, Gebrian B, St Jean R, Katz RV. Effect of childhood malnutrition on salivary flow and pH. Arch Oral Biol. 2008 Mar;53(3):231-7. doi: 10.1016/j.archoralbio.2007.09.007. Epub 2007 Nov 5. PMID 17983611
- [Background] Reddy V, Raghuramulu N, Bhaskaram C. Secretory IgA in protein-calorie malnutrition. Arch Dis Child. 1976 Nov;51(11):871-4. doi: 10.1136/adc.51.11.871. PMID 827242
- [Background] Rodriguez PN, Martinez Reinoso J, Gamba CA, Salgado PA, Mateo MT, Manto Mdel C, Molgatini SL, Iglesias V, Argentieri AB. Association among salivary flow rate, caries risk and nutritional status in pre-schoolers. Acta Odontol Latinoam. 2015;28(2):185-91. doi: 10.1590/S1852-48342015000200015. PMID 26355891
- [Background] Simoes A, de Campos L, de Souza DN, de Matos JA, Freitas PM, Nicolau J. Laser phototherapy as topical prophylaxis against radiation-induced xerostomia. Photomed Laser Surg. 2010 Jun;28(3):357-63. doi: 10.1089/pho.2009.2486. PMID 19814701
- [Derived] Vieira KA, Bastos CM, Vitor MGC, Deana AM, Fernandes KPS, Rodrigues MFSD, Pavesi VCS, Bussadori SK. Use of low-level laser therapy on children aged 1 to 5 years with energy-protein malnutrition: A clinical trial. Medicine (Baltimore). 2018 Apr;97(17):e0538. doi: 10.1097/MD.0000000000010538. PMID 29703031